CLINICAL TRIAL: NCT03833219
Title: Comparative Effectiveness of Financial Incentives and Smartphone-based Nudges to Reduce Cellphone Use While Driving Among Auto Insurance Policy Holders With Usage Based Insurance Policies
Brief Title: Comparative Effectiveness of Financial Incentives and Nudges to Reduce Cellphone Use While Driving Among UBI Auto Policy Holders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: U.S. Department of Transportation Federal Highway Administration (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 693JJ31750012
Record Dates: First submitted 2018-09-07; First posted 2019-02-06 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Automobile Accident
Keywords: distracted driving automobile; behavioral economics; usage-based insurance; auto insurance; automobile; smartphone application

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Control (monitor only) (No Intervention): Continue in monitoring only mode
- Social comparison feedback (Experimental): Report user's handheld phone use/ hour of driving for week. Compare this week's performance to distribution for driver cohort.
  Interventions: Behavioral: Weekly feedback
- End of rating period incentive (Experimental): Monitor throughout intervention period and compare overall use to distribution for cohort. Notify participant at end of intervention period regarding the amount they have earned.
  Interventions: Behavioral: End of intervention period incentive
- End of rating period incentive + social comparison feedback (Experimental): Monitor throughout intervention period and compare weekly phone use to driver cohort distribution. Send weekly push notification to provide feedback. Notify participant at end of intervention period regarding the amount they have earned.
  Interventions: Behavioral: Weekly feedback; Behavioral: End of intervention period incentive
- Weekly loss-framed incentive + social comparison feedback (Experimental): Monitor throughout intervention period and compare weekly phone use to driver cohort distribution. Send weekly push notification to provide feedback. Notify participant weekly regarding the amount they have earned.
  Interventions: Behavioral: Weekly feedback; Behavioral: Loss-framed weekly incentive
- Larger weekly loss-framed incentive+social comparison feedback (Experimental): Monitor throughout intervention period and compare weekly phone use to driver cohort distribution. Send weekly push notification to provide feedback. Notify participant weekly regarding the amount they have earned. Incentive amount is higher than "Weekly loss-framed incentive + social comparison feedback" Arm.
  Interventions: Behavioral: Weekly feedback; Behavioral: Loss-framed weekly incentive

INTERVENTIONS:
Behavioral: Weekly feedback — Send push notification reporting user's handheld phone use while driving compared to distribution for driver cohort (age, geographic area) each week.
  Arms: End of rating period incentive + social comparison feedback; Larger weekly loss-framed incentive+social comparison feedback; Social comparison feedback; Weekly loss-framed incentive + social comparison feedback
Behavioral: End of intervention period incentive — Notify participant about potential incentive at the end of the intervention period, but do not provide weekly feedback about performance.
  Arms: End of rating period incentive; End of rating period incentive + social comparison feedback
Behavioral: Loss-framed weekly incentive — Send push notification reporting user's handheld phone use while driving compared to distribution for driver cohort (age, geographic area) each week. Pay participant weekly according to where they fall on the distribution each week.
  Arms: Larger weekly loss-framed incentive+social comparison feedback; Weekly loss-framed incentive + social comparison feedback

SUMMARY:
The investigators are proposing an experiment to help a national auto insurance company test behavioral economic strategies to reduce the amount of time policy holders actively use their cell phone while driving. Interventions include financial incentives, social comparison, and nudges, and survey data will also be collected. Data collected from this internal trial will be shared with the Penn research team and analyzed

ELIGIBILITY:
Inclusion Criteria:

* Progressive Snapshot Users with policy activated within recruitment period
* Progressive Snapshot policy holder in one of the following states and regions: MI, PA, TX, FL, TN, OR, GA, NE, OK, OH, MT, MO, NV, CT, WI, MD, KY, MN, NH, NJ, AZ, ME, LA, SC, CO, MS, IN, IA, AL, ND, UT, RI, WV, WY, IL, AR, DE, KS, SD, NM, VT, ID, and the District of Columbia
* Has an email address

Exclusion Criteria:

* Progressive Snapshot Mobile App not updated to enable push notifications
* Customer's residential address is in a state in which phone use while driving is factored into insurance rating
* Customer's Snapshot Mobile App does not collect trip data with all sensors active
* Customer in Snapshot program for < 30 days or more > 70 days

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2108 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Seconds of active phone use per hour of driving | 150 days
  Percentage of driving time engaging in active handheld phone use (also measured as seconds of distracted driving/hour of driving)

SECONDARY OUTCOMES:
Seconds of passive phone use per hour of driving | 150 days
  Seconds of passive handheld, non-call use per hour of driving
Hard breaking events per 100 miles | 150 days
  notifications turned off, drop out of study, app uninstall
Hard acceleration events per 100 miles | 150 days
  Hard acceleration events per 100 miles

CONTACTS AND LOCATIONS:
Overall Officials: M. Kit Delgado, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
PI will not own individual participant data

REFERENCES:
- [Background] Delgado MK, Wanner KJ, McDonald C. Adolescent Cellphone Use While Driving: An Overview of the Literature and Promising Future Directions for Prevention. Media Commun. 2016 Jun 16;4(3):79-89. doi: 10.17645/mac.v4i3.536. PMID 27695663
- [Background] French B, Small DS, Novak J, Saulsgiver KA, Harhay MO, Asch DA, Volpp KG, Halpern SD. Preference-adaptive randomization in comparative effectiveness studies. Trials. 2015 Mar 18;16:99. doi: 10.1186/s13063-015-0592-6. PMID 25887045
- [Background] Halpern SD, Ubel PA, Asch DA. Harnessing the power of default options to improve health care. N Engl J Med. 2007 Sep 27;357(13):1340-4. doi: 10.1056/NEJMsb071595. No abstract available. PMID 17898105
- [Background] Halpern SD, French B, Small DS, Saulsgiver K, Harhay MO, Audrain-McGovern J, Loewenstein G, Brennan TA, Asch DA, Volpp KG. Randomized trial of four financial-incentive programs for smoking cessation. N Engl J Med. 2015 May 28;372(22):2108-17. doi: 10.1056/NEJMoa1414293. Epub 2015 May 13. PMID 25970009
- [Background] Hayashi Y, Russo CT, Wirth O. Texting while driving as impulsive choice: A behavioral economic analysis. Accid Anal Prev. 2015 Oct;83:182-9. doi: 10.1016/j.aap.2015.07.025. Epub 2015 Aug 13. PMID 26280804
- [Background] Klauer SG, Guo F, Simons-Morton BG, Ouimet MC, Lee SE, Dingus TA. Distracted driving and risk of road crashes among novice and experienced drivers. N Engl J Med. 2014 Jan 2;370(1):54-9. doi: 10.1056/NEJMsa1204142. PMID 24382065
- [Background] Lahrmann H, Agerholm N, Tradisauskas N, Berthelsen KK, Harms L. Pay as You Speed, ISA with incentive for not speeding: results and interpretation of speed data. Accid Anal Prev. 2012 Sep;48:17-28. doi: 10.1016/j.aap.2011.03.015. Epub 2011 Apr 9. PMID 22664664
- [Background] Loewenstein G, Brennan T, Volpp KG. Asymmetric paternalism to improve health behaviors. JAMA. 2007 Nov 28;298(20):2415-7. doi: 10.1001/jama.298.20.2415. No abstract available. PMID 18042920
- [Background] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Eberbach K, Walters KJ, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Individual Versus Team-Based Financial Incentives to Increase Physical Activity: A Randomized, Controlled Trial. J Gen Intern Med. 2016 Jul;31(7):746-54. doi: 10.1007/s11606-016-3627-0. Epub 2016 Mar 14. PMID 26976287
- [Background] Reagan IJ, Bliss JP, Van Houten R, Hilton BW. The effects of external motivation and real-time automated feedback on speeding behavior in a naturalistic setting. Hum Factors. 2013 Feb;55(1):218-30. doi: 10.1177/0018720812447812. PMID 23516803
- [Derived] Delgado MK, Ebert JP, Xiong RA, Winston FK, McDonald CC, Rosin RM, Volpp KG, Barnett IJ, Small DS, Wiebe DJ, Abdel-Rahman D, Hemmons JE, Finegold R, Kotrc B, Radford E, Fisher WJ, Gaba KL, Everett WC, Halpern SD. Feedback and Financial Incentives for Reducing Cell Phone Use While Driving: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2420218. doi: 10.1001/jamanetworkopen.2024.20218. PMID 38985474
- See also: Center for Insurance Policy Research. Usage-Based Insurance and Telematics. National Association of Insurance Commissioners. — http://www.naic.org/cipr_topics/topic_usage_based_insurance.htm
- See also: State Farm. (2014). Distracted Driving — http://teendriving.statefarm.com/road-to-safety/risky-driving/distracted-driving

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/19/NCT03833219/Prot_SAP_001.pdf